CLINICAL TRIAL: NCT07093957
Title: Effect of Delivery Method on Umbilical Cord Metabolomic Analysis
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ekin Guran, MD, Anesthesiologist, Aksaray University Training and Research Hospital
Other Study IDs: CORD_omics
Record Dates: First submitted 2025-07-17; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Metabolomics; Cord Blood
Keywords: cord blood; metabolomics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — Cord blood metabolome analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- C/S: Babies delivered via C/S
- Vaginal: Babies delivered vaginally

SUMMARY:
Birth type is closely linked to fetal and maternal stress responses. In this study, we aimed to examine the effects of delivery method on the stress response in newborns at the metabolite level.

DETAILED DESCRIPTION:
Birth type is closely linked to fetal and maternal stress responses. Previous studies have found higher levels of hormones associated with stress responses in mothers who delivered vaginally compared to those who delivered by cesarean section (C/S). Similarly, differences in markers assessing stress responses in newborns have been observed based on delivery method. However, the literature lacks sufficient studies on low-molecular-weight metabolites, which reveal the metabolic status of newborns.

Metabolomic profiling studies are introductory studies that provide comprehensive information about cell or organism metabolism. They contribute to research in many areas of medicine. In perinatology, metabolomic profiling studies have been conducted on topics such as neural tube defects, intrauterine growth restriction, and maternal diabetes. In this study, we aimed to examine the effects of delivery method on the stress response in newborns at the metabolite level.

ELIGIBILITY:
Inclusion Criteria:

* 1) Female patient aged 18-35 2) Term pregnancy 3) Pregnant with follow-up

Exclusion Criteria:

* 1) Having been diagnosed with diabetes mellitus before or during pregnancy 2) Having been diagnosed with hypertension before or during pregnancy 3) Non-singleton pregnancy 4) Non-elective C/S 5) Fetal intrauterine growth restriction 6) Mothers and their babies with a fetal birth anomaly or suspected birth anomaly will not be included in this study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population included pregnant women aged between 18 and 35 years who were regularly followed during their pregnancy and delivered at term. Women with a diagnosis of diabetes mellitus or hypertension either before or during pregnancy were excluded from the study. Additionally, pregnancies with multiple fetuses, non-elective cesarean sections, intrauterine growth restriction, or fetal congenital anomalies (or suspicion thereof) were not included. The study aimed to ensure a homogeneous and healthy sample to evaluate neonatal stress responses in relation to the mode of delivery.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
cord blood metabolomic analysis | From enrollment to birth. Cord Blood is taken during birth
  Cord blood samples will be analysed via LC/MS analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Huang Y, Ni Y, Meng Y, Zeng X, He X, Zhang L, Zhang J. Integrated proteomics and metabolomics network analysis across different delivery modes in human pregnancy: a pilot study. BMC Pregnancy Childbirth. 2024 Dec 26;24(1):868. doi: 10.1186/s12884-024-07097-4. PMID 39725908
- [Background] Shokry E, Marchioro L, Uhl O, Bermudez MG, Garcia-Santos JA, Segura MT, Campoy C, Koletzko B. Investigation of the impact of birth by cesarean section on fetal and maternal metabolism. Arch Gynecol Obstet. 2019 Sep;300(3):589-600. doi: 10.1007/s00404-019-05213-w. Epub 2019 Jun 14. PMID 31201538
- [Background] Ross AB, Barman M, Hartvigsson O, Lundell AC, Savolainen O, Hesselmar B, Wold AE, Sandberg AS. Umbilical cord blood metabolome differs in relation to delivery mode, birth order and sex, maternal diet and possibly future allergy development in rural children. PLoS One. 2021 Jan 25;16(1):e0242978. doi: 10.1371/journal.pone.0242978. eCollection 2021. PMID 33493154